CLINICAL TRIAL: NCT06166394
Title: Pharmacodynamic Profile of Intrathecal Hypobaric Local Anesthetics. An Observational Study
Brief Title: Spinal Hypobaric Local Anesthetic Study
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5558; v04Nov2022 (Other: UHN)
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia, Local
Keywords: Spinal Hypobaric LA; Bupivacaine; Mepivacaine
MeSH Terms: interventions — Mepivacaine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mepivacaine: Day surgery patients(30 patients); For these patients- Administration of a spinal hypobaric mepivacaine injection
  Interventions: Drug: Spinal hypobaric Mepivacaine Local Anesthetic Injection
- Bupivacaine: In-patients(30 patients): For these patients- Administration of a spinal hypobaric bupivacaine injection
  Interventions: Drug: Spinal hypobaric Bupivacaine Local Anesthetic Injection

INTERVENTIONS:
Drug: Spinal hypobaric Mepivacaine Local Anesthetic Injection — • Administration of a hypobaric spinal mixture for Day-Surgery patients: 3.4ml of 1.5% mepivacaine created by 3ml 2% mepivacaine with 1ml sterile water, and then discarding 0.6ml
  Other Names: Carbocaine
  Groups: Mepivacaine
Drug: Spinal hypobaric Bupivacaine Local Anesthetic Injection — Administration of a hypobaric spinal mixture for In-patients:
  3ml of 0.33% bupivacaine created by 2ml 0.5% bupivacaine with 1ml sterile water
  Other Names: Marcaine
  Groups: Bupivacaine

SUMMARY:
The length of hospital stay after total hip and knee arthroplasty is determined based on the successful mobilization of the patients post surgery. Fast track pathways involving early mobilization and discharge of the patient on the same day of surgery, shortens the hospital stay and reduces the risk of adverse effects. The long acting LA (bupivacaine) is most commonly used in spinal anesthesia for arthroplasty surgeries and is associated with a prolonged motor and sensory block. In contrast, hypobaric bupivacaine and hypobaric mepivacaine helps in achieving the desired block level with smaller dosage and shorter onset time and faster recovery when compared to long acting local anesthetics. The aim of the study is to observe the effects of hypobaric local anesthetics ( bupivacaine and mepivacaine ) in patients undergoing unilateral total hip or knee arthroplasty in terms of time to onset and time to recovery of the block and also its effect on hemodynamic stability and time to mobilization after surgery. This study will allow the investigators to recommend optimal dosing strategies that in turn will help in faster recovery from spinal anesthesia and early mobilization thereby reducing harmful outcomes.

DETAILED DESCRIPTION:
Fast-track pathways involving same day mobilization and hospital discharge for total hip and knee arthroplasty are increasingly popular in modern orthopedic practice. Numerous reports have demonstrated the feasibility of this approach.

The choice of local anesthetic (LA) drug and dose administered in spinal anesthesia is determined by several considerations including the desired block height (the upper limit of sensory loss and surgical anesthesia that is achieved) and block duration. Block height and duration should be adequate for the surgery in question, but should ideally not be excessive, as they can lead to adverse effects including sympathetic blockade and hypotension, urinary retention, and delayed recovery of motor function in the lower limbs. The long-acting amide LA, bupivacaine, is most commonly used in this setting at Toronto Western Hospital (TWH) and elsewhere in the world. It is, however, associated with a prolonged motor and sensory recovery (4-6 hours). An alternative strategy to achieve adequate block height without using excessive doses of LA is to administer a hypobaric solution of bupivacaine or mepivacaine; this has been trialed with success at TWH and is now used routinely by staff anesthesiologists. Nevertheless, most of the investigator's knowledge regarding hypobaric LA solutions in spinal anesthesia comes from studies that are more than two decades old. There are no studies on mepivacaine, and neither hypobaric bupivacaine nor mepivacaine have been investigated in the context of fast-track total hip and knee arthroplasty pathways. In this context, the ideal LA solution used for spinal anesthesia should provide a consistent and fast onset time to achieve the required surgical anesthesia while the sensory and motor block should resolve as soon as possible after surgery. The investigators believe that hypobaric bupivacaine and hypobaric mepivacaine may satisfy these criteria and hence, the investigators aim to study their pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective unilateral total hip or knee arthroplasty under spinal anesthesia at Toronto Western Hospital
2. American Society of Anesthesiologists physical status class (ASA-PS) 1-3
3. Aged ≥ 20 years

Exclusion Criteria:

1. Refusal to participate
2. Inability to communicate due to language barrier or cognitive impairment
3. Height < 150 cm or > 200 cm
4. Weight < 40 kg or >130 kg
5. Contraindication or allergy to amide-type local anesthetic
6. Contraindication to spinal anesthesia (e.g., infection at the injection site, existing coagulopathy)
7. Spinal anesthesia performed in the operating room rather than the block room (which will preclude adequate testing)
8. Spinal anesthesia that includes administration of intrathecal opioids (e.g., morphine, fentanyl),so as to avoid unanticipated alterations in block quality or solution baricities.
9. Pre-existing sensory or motor impairment in the lower extremities

   -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All day surgery and in-patients who are scheduled to undergo elective unilateral total hip or knee arthroplasty under spinal anesthesia at Toronto Western Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
1. Time to reach the most cephalad/cranial sensory block level (onset time of spinal anesthesia on the surgical side). | Assessed over the duration of time period till the patient is discharged.
  Time to onset is a continuous variable and therefore will be expressed as mean ± standard deviation.
Time to reach sensory block level of L1 or higher (adequate level of anesthesia for knee surgery) on the surgical side | Assessed over the duration of time period till the patient is discharged.
  Time to onset is a continuous variable and therefore will be expressed as mean ± standard deviation.
Time to reach sensory block level T10 or higher (adequate level of anesthesia for hip surgery) on the surgical side | Assessed over the duration of time period till the patient is discharged.
  Time to onset is a continuous variable and therefore will be expressed as mean ± standard deviation.
The most cephalad/cranial sensory block level | Assessed over the duration of time period till the patient is discharged.
  Sensory block will be assessed every 5 mins during the first 30 mins after spinal injection. A pinprick test using an 18G (Gauge) blunt-tipped needle (BD Blunt Fill needle) will be performed on non-dependent and dependent sides to detect sensory loss over the torso and lower limbs.
Time to achieve complete motor block on the modified Bromage scale | Assessed over the duration of time period till the patient is discharged.
  Time to onset is a continuous variable and therefore will be expressed as mean ± standard deviation.

SECONDARY OUTCOMES:
Time to regression of the sensory block to the L2 dermatome on both lower limbs. | Assessed over the duration of time period till the patient is discharged.
  Time to onset is a continuous variable and therefore will be expressed as mean ± standard deviation.
Time to full motor recovery on the modified Bromage scale | Assessed over the duration of time period till the patient is discharged.
  Time to onset is a continuous variable and therefore will be expressed as mean ± standard deviation.
Hemodynamic stability after the spinal injection | Assessed over the duration of time period till the patient is discharged.
  Will be assessed by the measurement of vitals
Time to ambulation | Assessed over the duration of time period till the patient is discharged.
  Time to onset is a continuous variable and therefore will be expressed as mean ± standard deviation.
Patient satisfaction score | Assessed before the patient is discharged.
  Assessed by a five-point Likert scale provided to the patient
Surgeon's perception of quality of anesthesia | Assessed after the end of surgery.
  Assessed by a three-point Likert scale provided to the surgeon
Rate of successful spinal anesthesia | Assessed after the spinal block till the end of surgery
  Will be determined as successful when there will be no need to convert to general anesthesia or administer supplemental opioids or local infiltration in the operating room.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jinn Chin, MD,FRCPC, Principal Investigator — UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No